CLINICAL TRIAL: NCT06586515
Title: A Phase 1a/1b Trial of LY3962673 in Participants With KRAS G12D-Mutant Solid Tumors
Brief Title: MOONRAY-01, A Study of LY3962673 in Participants With KRAS G12D-Mutant Solid Tumors
Acronym: MOONRAY-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27189; J5J-OX-JZZA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non-small Cell Lung Cancer; Colorectal Cancer
Keywords: KRAS G12D; KRAS; LY3962673; Cetuximab; nab-paclitaxel; Gemcitabine; Oxaliplatin; Leucovorin; Irinotecan; 5-fluorouracil
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — Cetuximab; Gemcitabine; 130-nm albumin-bound paclitaxel; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Phase 1a/1b
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a: LY3962673 Dose Escalation (Experimental): Escalating doses of LY3962673 administered orally.
  Interventions: Drug: LY3962673
- Phase 1b: LY3962673 Dose Expansion (Experimental): LY3962673 administered orally either alone or in combination with other chemotherapy agents.
  Interventions: Drug: LY3962673; Drug: Cetuximab; Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: Oxaliplatin; Drug: leucovorin; Drug: Irinotecan; Drug: 5-fluorouracil
- Experimental: Phase 1a: LY3962673 Monotherapy (Experimental): LY3962673 administered orally
  Interventions: Drug: LY3962673

INTERVENTIONS:
Drug: LY3962673 — Administered orally.
Drug: Cetuximab — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion
Drug: Gemcitabine — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion
Drug: nab-paclitaxel — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion
Drug: Oxaliplatin — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion
Drug: leucovorin — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion
Drug: Irinotecan — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion
Drug: 5-fluorouracil — Administered intravenously.
  Arms: Phase 1b: LY3962673 Dose Expansion

SUMMARY:
The main purpose of this study is to assess safety & tolerability and antitumor activity of LY3962673 as monotherapy and in combination with other chemotherapy agents in participants with KRAS G12D-mutant advanced solid tumor types. The study is expected to last approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have Histological or cytologically proven diagnosis of locally advanced, unresectable, and/or metastatic cancer and measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Have evidence of KRAS G12D mutation in tumor tissue or circulating tumor DNA
* Have an ECOG performance status of ≤ 1
* Must have received ≥ 1 prior line of systemic chemotherapy for advanced or metastatic disease
* Participants with asymptomatic or treated CNS disease may be eligible.

Exclusion Criteria:

* Have known active CNS metastases and/or carcinomatous meningitis.
* Have any unresolved toxicities from prior therapy greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 1.
* Have significant cardiovascular disease as unstable angina or acute coronary syndrome, history of myocardial infarction, known reduced left ventricular ejection fraction.
* Have active uncontrolled systemic bacterial, viral, fungal, or parasitic infection.
* Have known active hepatitis B virus (HBV) and hepatitis C virus (HCV).
* Have other active malignancy unless in remission with life expectancy greater than (>) 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through 5 years
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.
Phase 1a: Number of Participants with DLT | During the first 28-day cycle of LY3962673 treatment
Phase 1a: Number of Participants with DLT Equivalent Toxicities | During the first 28-day cycle of LY3962673 treatment
Phase 1b: Overall Response Rate (ORR) | Up to approximately 5 years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Phase 1b: Best Overall Response (BOR) | Up to approximately 5 years
  BOR per investigator assessed RECIST 1.1
Phase 1b: Duration of Response (DOR) | Up to approximately 5 years
  DOR per investigator assessed RECIST 1.1
Phase 1b: Time to Response (TTR) | Up to approximately 5 years
  TTR per investigator assessed RECIST 1.1
Phase 1b: Disease Control Rate (DCR) | Up to approximately 5 years
  DCR per investigator assessed RECIST 1.1

SECONDARY OUTCOMES:
Phase 1a: Overall Response Rate (ORR) | Up to approximately 5 years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Best Overall Response (BOR) | Up to approximately 5 years
  BOR per investigator assessed RECIST 1.1
Duration of Response (DOR) | Up to approximately 5 years
  DOR per investigator assessed RECIST 1.1
Time to Response (TTR) | Up to approximately 5 years
  TTR per investigator assessed RECIST 1.1
Disease Control Rate (DCR) | Up to approximately 5 years
  DCR per investigator assessed RECIST 1.1
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3962673 | Predose through Day 168
  PK: Cmax of LY3962673
PK: Time to Maximum Concentration (Tmax) of LY3962673 | Predose through Day 168
  PK: Tmax of LY3962673
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3962673 | Predose through Day 168
  PK: AUC of LY3962673

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- United States (25):
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Lake Nona - Sarah Cannon Research Institute, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Community Health Network, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - New York University (NYU) Langone Medical Center, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati (UC) - Cancer Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - USO - US Oncology Research Network, Nashville, Tennessee
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
- Canada (2):
  - The Ottawa Hospital, Ottawa
  - Princess Margaret Hospital, Toronto
- China (4):
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing
  - Beijing Cancer hospital, Beijing
  - Harbin Medical University Cancer Hospita, Harbin
  - Fudan University Cancer Center, Shanghai
- France (4):
  - Centre Leon Berard, Lyon
  - Centre d'Essais Precoces en Cancerologie de Marseille (CEPCM) - AP-HM Hopital de La Timone, Marseille
  - Oncopole Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München
- START Dublin Early Phase Clinical Trials Unit, Dublin, Ireland
- Italy (3):
  - Azienda Ospedaliera Universitaria - Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - UOC Fase I - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Roma
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Japan (5):
  - National Cancer Center Hospital East, Chiba
  - Kanagawa cancer center, Kanagawa
  - Aichi Cancer Center Hospital, Nagoya
  - Kansai Medical University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
- Spain (4):
  - South Texas Accelerated Research Therapeutics (START) Barcelona- HM Nou Delfos, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3962673 in Participants With KRAS G12D-Mutant Solid Tumors — https://trials.lilly.com/en-US/trial/533076